CLINICAL TRIAL: NCT05681364
Title: Prediction of Pulmonary Rehabilitation Outcomes in Patients With Chronic Respiratory Disease Based on Metabolomics: a Prospective Cohort Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 01
Record Dates: First submitted 2022-10-19; First posted 2023-01-12 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2022-10

CONDITIONS: Chronic Obstructive Pulmonary Disease; Bronchiectasis
Keywords: pulmonary rehabilitation; chronic respiratory disease; metabonomics
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum and exhaled breath condensate
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COPD and bronchiectasis patients with some metabolic profiling: The patients with stable COPD and bronchiectasis who meet the screening criteria and with some metabolic profiling according to the previous studies.
  Interventions: Other: metabonomics
- COPD and bronchiectasis patients without the metabolic profiling: The patients with stable COPD and bronchiectasis who meet the screening criteria and without the metabolic profiling according to the previous studies.
  Interventions: Other: metabonomics

INTERVENTIONS:
Other: metabonomics — profiles of metabolites in serum and exhale breath condensate (EBC) at baseline and after pulmonary rehabilitation

SUMMARY:
To comprehensively evaluate the pulmonary rehabilitation (PR) outcomes of patients with chronic respiratory disease (CRD), and to screen biomarkers for predicting different PR outcomes of patients with CRD using metabolomics methods, and to build a prediction model.

ELIGIBILITY:
Inclusion Criteria:

* For COPD

  1. Meets the Global initiative for chronic obstructive lung disease (GOLD) 2022 definition of stable COPD;
  2. Age 30-75 years;
  3. Lung CT images only showed chronic bronchitis and emphysema;
  4. Agree to participate in the study and is able to cooperate with exhaled breath condensate collection.
* For bronchiectasis

  1. Lung CT showed bronchiectasis;
  2. Age 18-75 years;
  3. Spirometry suggests obstructive ventilatory dysfunction: forced expiratory volume in one second (FEV1) is less than 70% of forced vital capacity (FVC) post bronchodilator inhalation.

Exclusion Criteria:

1. Asthma or other respiratory diseases
2. History of pulmonary surgery
3. α1 antitrypsin deficiency
4. Autoimmune diseases
5. Patients with acute myocardial infarction, chronic heart failure, severe cerebral infarction or cerebral hemorrhage
6. A history of malignant disease now or within 2 years
7. History of acute exacerbation or change of medication in the past 4 weeks
8. A history of blood transfusion within the last 4 weeks
9. Drugs or alcohol abuse
10. Breastfeeding or pregnant women
11. Unable to cooperate with pulmonary rehabilitation for various reasons

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients in respiratory and critical care medicine department of Peking University Third Hospital
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pulmonary rehabilitation outcome | At week 12 of pulmonary rehabilitation
  Systemic multidimensional measurements （SMM） will be used to evaluate the outcomes of PR program, the patients will be grouped in very good, good, moderate and poor responders by cluster analysis.
  SMM are as follows: changes in the degree of dyspnea will be measured using the modified Medical Research Council scale; the St George's Respiratory Questionnaire will be use to evaluate changes in health status; exercise performance will be measured by a 6-min walk test and a constant work-rate test; the Canadian Occupational Performance Measure will be used to identify specific problematic activities of daily life; patients scored how well they were performing the problematic activities of daily life and how satisfied they were with this level of performance; symptoms of anxiety and depression will be measured by Hospital Anxiety and Depression Scale. The efficacy of the PR program of the whole sample will be evaluated based on the minimal clinically importance.

CONTACTS AND LOCATIONS:
Overall Officials: Fei Wang, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: Undecided